CLINICAL TRIAL: NCT02172209
Title: The Effect of Food on the Bioavailability and Pharmacokinetics of BI 10773 Tablet, Administered as a Single Dose of 50 mg With and Without Food to Healthy Male Volunteers in an Open-label, Randomised Intraindividual Crossover Comparison Design
Brief Title: Bioavailability and Pharmacokinetics of BI 10773 Tablet in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1245.3
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — empagliflozin

ARMS (2):
- BI 10773 tablet administered with food (Experimental): 50 mg BI 10773 after a standardised high fat breakfast
  Interventions: Drug: BI 10773
- BI 10773 tablet administered to fasted subjects (Active Comparator): 50 mg BI 10773 p.o. after an overnight fast of at least 10 hours
  Interventions: Drug: BI 10773

INTERVENTIONS:
Drug: BI 10773

SUMMARY:
Trial to assess the effect of food on the pharmacokinetics and the extent of absorption of a single dose BI 10773 tablet in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy males according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (BP, HR), 12-lead ECG, clinical laboratory tests
* Age ≥ 18 and Age ≤ 55 years
* BMI ≥ 18.5 and BMI ≤ 29.9 kg/m2
* Signed and dated written informed consent prior to admission to the study in accordance with GCP (Good Clinical Practice) and the local legislation

Exclusion Criteria:

* Any finding in the medical examination (including BP (blood pressure), PR (pulse rate) and ECG (electrocardiogram)) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with the dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g. repeated demonstration of a QTc interval >450 MS)
* A history of additional risk factors for torsade de pointes (e.g. heart failure, hypokalemia, family history of Long QT Syndrome)
* Elevated urinary glucose levels at screening (> 15 mg/dl; > 0.83 mmol/L)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2008-01; Primary Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 hours post dose
Cmax (maximum measured concentration of the analyte in plasma) | Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 hours post dose

SECONDARY OUTCOMES:
tmax (time from dosing to the maximum concentration of the analyte in plasma) | Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 hours post dose
t1/2 (terminal half-life of the analyte in plasma) | Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 hours after last dose
%AUCtz-∞ (the percentage of the AUC0-∞ that is obtained by extrapolation) | Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 hours post dose
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 hours post dose
λz (terminal rate constant in plasma) | Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 hours post dose
MRTpo (mean residence time of the analyte in the body after p.o. administration) | Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 hours post dose
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 hours post dose
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 hours post dose
Glucose excretion in urine | pre-dose and 0-4, 4-8, 8-12, 12-24 hours post-dose
Creatinine excretion in urine | pre-dose and 0-4, 4-8, 8-12, 12-24 hours post-dose
Abnormal findings in physical examination | Baseline and within 14 days after last trial procedure
Changes from baseline in vital signs (blood pressure, pulse rate) | Baseline and within 14 days after last trial procedure
Changes from baseline in 12-lead ECG (electrocardiogram) | Baseline and within 14 days after last trial procedure
Changes from baseline in routine laboratory tests | Baseline and within 14 days after last trial procedure
Incidence of adverse events | Up to 15 days
Assessment of tolerability by investigator on a 4-point scale | Within 14 days after last trial procedure